CLINICAL TRIAL: NCT05193578
Title: Home-based Intervention With Semaglutide Treatment Of Neuroleptica-Related Prediabetes
Acronym: HISTORI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jan Frystyk (Other)
Collaborators: Region Zealand (Other); Region of Southern Denmark (Other); Steno Diabetes Center Sjaelland (Other Government); Steno Diabetes Center Odense (Other)
Responsible Party: Sponsor-Investigator, Jan Frystyk, Professor, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Eudra CT 2020-004374-22
Record Dates: First submitted 2021-12-09; First posted 2022-01-18 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Schizophrenia; Prediabetic State
Keywords: Randomized Controlled Trial; Metabolic Syndrome; Overweight; Glucagon-Like Peptide 1; Cardiovascular Diseases; Positive and negative symptoms (PANSS); Quality of Life
MeSH Terms: conditions — Schizophrenia; Prediabetic State; Metabolic Syndrome; Overweight; Cardiovascular Diseases | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The un-blinding will occur after the data analysis have ended and two blinded conclusions have been uploaded to clinicaltrials.gov based on the results of the primary and secondary outcomes defined in the SAP. The two blinded conclusions are added to the SAP.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Semaglutide (Active Comparator): Active Comparator: Semaglutide injection once-weekly
  The participants start with Semaglutide given as 0.25 mg subcutaneously per week for 4 weeks. Then, the dose is uptitrated to 0.5 mg subcutaneously per week for 4 weeks, whereafter the highest dose is reached: 1 mg subcutaneously per week until the end of the study (week 30).
  Subjects, who experience side effects that hinder a stepwise increase in study drug, will remain at the highest possible tolerated dose for the rest of the study.
  Interventions: Drug: Semaglutide, 1.34 mg/mL
- Placebo (Placebo Comparator): Semaglutide-Placebo injections once weekly.
  The Semaglutide-Placebo pens are produced by Novo Nordisk A/S and resemble the pens containing active drug.
  Semaglutide-Placebo pens contain vehicle, i.e. no active drug. Semaglutide-Placebo is administered similarly to semaglutide. That is using the same uptitration regime and volume as the active comparator, Semaglutide.
  Subjects, who experience side effects that hinder a stepwise increase in Semaglutide-Placebo, will remain at the highest possible tolerated dose for the rest of the study.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Semaglutide, 1.34 mg/mL — Semaglutide, 1.34 mg/mL
  Arms: Semaglutide
Other: Placebo — Semaglutide-Placebo
  Arms: Placebo

SUMMARY:
To investigate whether the Glucagon Like Peptide 1 (GLP-1) Semaglutide (1.34 mg/ml) has preventive effect compared to placebo in the development of diabetes and Metabolic Syndrome in people with pre-diabetes, overweight and schizophrenia, who receive antipsychotic treatment.

Furthermore to investigate for an effect of Semaglutide compared to placebo on psychotic symptoms and quality of life in people with schizophrenia, prediabetes and overweight.

DETAILED DESCRIPTION:
Quality control:

Usual quality control procedures will be followed in accordance with the ICH Guideline for Good Clinical Practice (GCP). The GCP unit at OUH will be responsible for monitoring the study in accordance with GCP guidelines. This protocol will be submitted as part of the notification to the Danish Medicines Agency and the Scientific Ethical Committee for the Region of Southern Denmark. Data processing regarding the trial will be reported to the Region's list of on-going research projects via the Executive Secretariat at OUH. Furthermore, Novo Nordisk will be informed of the trial.

Randomization:

A total of 154 participants will be randomized: 77 participants will be randomized to the Semaglutide group and 77 participants will be randomized to the placebo group (randomization ratio 1:1). The participant is assigned a subject number when consent is obtained, inclusion and exclusion criteria have been reviewed and the participant otherwise meets the requirements for study participation and continues to participate in the study. A participant cannot be assigned more than one randomization number and this number cannot be used for other persons. Block randomization including blocks of either 4 or 6 randomization numbers will be used, and the randomisations list will be provided by the manufacturer of Semaglutide and placebo (Novo Nordisk). The randomization will take place via the RedCAP® module.

Treatment arm allocation will be concealed to investigators. Randomization codes will be delivered in closed envelopes, kept in Odense, Denmark, in a secure place with 24-hour access.

Novo Nordisk A/S is going to provide the randomization list. The investigators of the trial are blinded and will randomize subjects via the Novo Nordisk provided blinded randomization list. Subsequently, the investigators inform the unblinded staff not otherwise involved in the trial. The staff is then using the unblinded version of the randomization list to identify the treatment arm that this specific patient is randomized to. Then, the staff allocates the correct trial product via a unique dispensing number (DUN) on the box and on an unblinded total DUN list.

Biological material / biobank:

Biological material will be stored in a research biobank to be analysed at the end of trial.

In addition biological material will also be collected and stored in a biobank for future research projects. Biological material will be stored in pseudo-anonymised form by ID-number in a biobank for 15 years, after which it will be destroyed. In case there is a need for further studies of biomaterial, application will again be made to the local Scientific Ethical Committee.

Data management:

Data from the trial will be stored with the data controller. The study's data processing will be reported to the Region of Southern Denmark's list of on-going research projects. All data will be available to co-authors of any articles based on the study, and data will also be available to the journals or authorities that may have a legitimate interest in accessing the data. In addition, data will be available for monitoring of project as the investigator allows direct access to source data/documents (including patient medical records) for monitoring, auditing and/or inspection by the GCP units, the Danish Medicines Agency and other countries' health authorities. There will be a collaboration with OPEN (Open Patient data Explorative Network, Odense, Denmark) in order to receive help to use and manage RedCAP®. Source data will be entered into or transferred to the RedCAP® module, and scan documents will be archived as source documents. All transferred documents to RedCAP® will be archived for five years after the end of the trial, after which they will be destroyed. Source data in the form of patient medical records will be handled by Odense University Hospital.

Recruitment:

To embed the study in the community psychiatry centers teams, the investigators need help from local consultants in psychiatry. Their task is to help to identify and enroll patients.

If a potential participant is interested in obtaining more information regarding the trial, the potential participant may contact the research units involved via phone or e-mail. An investigator or another member of the research staff (e.g. research technician or nurse) will contact the potential participant to answer upfront questions and to provide written information about the clinical trial.

By signing the informed consent, the participant gives permission to the Danish Medicines Agencies, Sponsor, investigator and monitor to have direct access to obtain information from the patient record including electronical records relevant for completion, surveillance or control of the clinical trial. All trial-related visits will take place in patients home or at the OPUS clinics and community psychiatry centers clinics in Region of southern Denmark or Zealand. The participants will be encouraged to bring an assessor to clinic visits.

Plan for participation:

Participation in the study will cease if the participant wishes to exit the study. Discontinuation may also occur at the investigators' request; for example, if a severe competing disorder or adverse side effects develop in the participant (up to a maximum of six weeks after the last scheduled injection), or if the participant is not compliant of the trial medication / placebo or in attendance for the administration of trial medication and the measurement of safety markers. The investigation may be terminated if information on new side effects emerges and, for this reason, the authorities recommend that the use of the medication cease. If a trial participant exits the study early, any provided biological material and scans will be included in the final analysis. If a trial participant withdraws the informed consent or exits the clinical trial before 30 weeks of treatment, no further analyses than those at the time point already planned and accepted by the participant, will be done on the biomaterial obtained from the participant. Unless the participant, who withdraws the informed consent or exits the clinical trial before 30 weeks of treatment specifically asks for destruction of the already obtained biological material, it will be stored in the biobank in accordance with the described precautions in this protocol. If more than 15% of the participants exit within three months of the start of the trial, they will be replaced by the inclusion of other participants. Patients withdrawing from the trial should be encouraged to undergo same final evaluation as patients completing trial.

eCRF: The purpose of CRF is to report all the information required by the protocol of the individual trial participants. Electronic CRF (eCRF) will be used. Completion of CRF will begin with the recruitment of the participants and filled in continuously throughout the trial by the investigators (or persons appointed by the investigators who are either experienced in using RedCAP® (or who will receive training prior to the assignment). CRF is the source document for trial data that is written directly into the eCRF and which is not first recorded in the Medical journal.

Source data, which is recorded directly in the eCRFs, includes protocol-specific measurements that are not relevant in the patient's medical record. eCRF is managed by the Odense Patient Data Explorative Network, SDU, Odense, using the RedCAP® system.

Effect analyses:

All participants randomized in the study will be included in the assessment of endpoints. Clinical results will be presented as mean, least squares mean, least square mean change from baseline or least square difference between groups with SE, SD or two-sided 95% CI. Statistical tests will be conducted as two-sided tests with a 5% significance level.

Primary outcomes for the study will be absolute changes in HbA1c. Changes in HbA1c will be evaluable after three months and after 6 months. A mixed effects linear regression analysis is used to compare changes in glucose tolerance, HbA1c, from baseline to six months' follow-up between the intervention and the placebo groups. Missing values will be imputed, primary analysis will be intention to treat. Supplementary per protocol analysis will accompany the intention to treat analysis.

The investigators conservatively assume that 6 months of semaglutide treatment changes HbA1c by 0.2%, and that SD equals 0.35%. Based on these assumptions, calculations show that 65 subjects in each arm are required to obtain a power of 90%, using a 2-sided significance level of 5%.

All changes in secondary outcomes from baseline to various follow-up times are analyzed using mixed effects linear regression analyses for continuous outcomes and mixed effects logistic regression analyses for categorical outcomes.

All analyses on continuous outcomes are adjusted for the baseline value of the outcome, and in case of large imbalances in baseline patient characteristics between the two randomized groups, exploratory analyses including such variables are conducted. To correct for multiple testing of the secondary outcomes, Holm's sequentially rejective multiple test procedure will be applied. Statistical analyses are performed using Stata software Version 16 (Statacorp, Texas, USA). The hypothesis tests are 2 sided, and the 5% level of significance is considered.

Safety:

At all visits, vital signs will be recorded, including blood pressure, body weight and waist circumference as well as adverse reactions, including information on possible cases of low blood sugar (hypoglycaemia). The safety parameters in the study include adverse reactions, vital parameters and biochemical studies (blood sugar as well as liver and kidney function). These parameters have been selected because they partly include the issues that the participant will have experienced (side effects) and partly the possible effects on vital functions, including blood pressure and liver and kidney function. Long-term blood sugar (HbA1c) and fasting blood sugar will be measured at attendance. When indicated, blood sugar will be measured by the study nurse on the regular visits. In theory, the drug can lower blood sugar, although it is only detected by concomitant treatment with other drugs to treat diabetes. If unrecognized illness is detected in participants - unless before the start of the study, they expressed a wish to the contrary - they will be informed of this and referred to the relevant healthcare professional or department. If any side effects or changes in biochemical anomalies are observed, the trial physician or the physician responsible for the test will be informed.

After 10 weeks of injections and given, that the study staff considers it safe, participants will be given the possibility to self-administer the injections under guidance via ether telephone or video.

All safety parameters will be recorded in the medical journal as soon as they have either been measured or reported by the test participant. The following information will be reported: Study name, patient identification including subject number and initials, sex and age, diagnosis, trial drug, causality assessment, outcome, and name of the reporter.

Publication of data:

All results, negative as well as positive, will be published in scientific journals and in EudraCT results database. Data will be transferred to the public data register after publication (www.clinicaltrials.gov), cf. agreement with the grant-awarding bodies that fund the investigation. ICMJE's author guidelines for scientific articles will be followed.

Funding:

Novo Nordisk Foundation. Steno Diabetes Center Zealand. Steno Diabetes Center Odense. Slagelsepuljen.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with schizophrenia spectrum disorder (ICD10 codes DF20, DF21 or DF25)
* Age between 18 and 60 years (both included)
* Approved contraception for female participants
* Treated by one of the OPUS clinics and or community psychiatry centers teams and community psychiatry in the Region of Southern Denmark or Zealand
* Antipsychotic SGA treatment for at least 6 months
* Stable co-medication for at least 1 month
* HbA1c between 39-47 mmol/mol (both included). Two measurements with ≥3 month interval are required to confirm prediabetes. The first measurement is identified and obtained from patient journals, the second prior to enrolment
* BMI ≥27 kg/m2. Two weights with ≥3 month interval are required to confirm obesity
* Capable of providing informed oral and written consent

Exclusion Criteria:

* Diagnosis of diabetes (T1D or T2D) or a HbA1c >47 mmol/mol
* Active malignant disease within the last 5 years
* Pregnancy or breast feeding
* Exceeding high risk consumption limit (>21 / 14 units of alcohol for men / women, respectively) or severe substance abuse
* Unwillingness to allow home visits by a study nurse
* Significant somatic disease: 1) end-stage renal failure (eGFR <15 ml/min); 2) elevated liver function tests (liver transaminases >2 times upper normal limit); 3) history of acute or chronic pancreatitis; 4) heart failure (NYHA class IV) or unstable angina pectoris or myocardial infarction with the last 6 months; 5) uncontrolled hypertension (systolic blood pressure >180 mm Hg, diastolic blood pressure >100 mm Hg)
* Previous treatment with study drug or use of other weight reducing drugs within the last 6 month
* Participation in other drug trials
* Treatment with drugs approved for overt diabetes type 2. (Metformin not included)
* Circumstances that the investigator believes will interfere with the trial

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 154 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
HbA1c (mmol/mol) | 30 weeks
  Absolute change in HbA1c reported as mmol/mol from baseline to end of treatment

SECONDARY OUTCOMES:
Weight | 30 weeks
  Absolute change in weight in kilogram
Height | 30 weeks
  Height measured in meters at baseline and after 30 weeks.
Chaneges in body mass index (BMI) | 30 weeks
  weight (kg) and height (meters) will be combined to report body mass index in kg/m^2 at baseline and after 30 weeks
Waist circumference (cm) | 30 weeks
  Absolute change in waist circumference as measured in cm by the study nurse
Glycemic status (blood sampling) | 30 weeks
  Absolute change in insulin resistance as estimated by HOMA, using fasting serum levels of insulin (measured in pmol/Liter) and plasma glucose (measured in mmol/Liter).
  HOMA is calculated using the formula provided by Matthews et al., 1985 in Diabetologia
Plasma triglyceride | 30 weeks
  Blood sample with plasma triglyceride (reported in mmol/Liter)
Cholesterol concentrations | 30 weeks
  Blood sample with cholesterol concentrations (reported in mmol/Liter)
Absolute change in systolic and diastolic blood pressure (mmHg) | 30 weeks
  Blood pressure is measured at home by study nurse while the participant is resting in a chair.
Cardiovascular risk markers | 30 Weeks
  Cardiovascular risk markers: cardiovascular autonomic neuropathy (CAN) (Vagus TM®), and circulating levels of cardiovascular risk markers. CAN is considered a serious complication of diabetes, being associated with a 5-fold increased risk of CVD. Of interest to this study, CAN may be present prior to the development of diabetes and it can be improved by weight loss. As CAN may be measured by a hand held apparatus (Vagus TM®), measurements are easily performed in the homes of the enrolled patients. CAN will be measured at inclusion, at 15 weeks and at end of study. Results will not be covered in primary publication. The results will be included in a publication decribing cardiovascular risk in study population.
Pro-atherosclerotic changes | 30 Weeks
  Pro-atherosclerotic changes: we want to perform a pilot study in a subsample of 20 participants from placebo vs. 20 participants from the Semaglutide group, focusing on pre-symptomatic atherosclerosis assessed by positron emission tomography/computed tomography (PET/CT) using 18F-sodium fluoride (NaF) as tracer. NaF-PET/CT is a novel way of detecting and measuring calcification in major arteries, potentially years or decades before manifest arterial wall calcification becomes detectable by cardiac CT. We plan to perform two NaFPET/CT acquisitions, i.e. at baseline and after 30 weeks treatment. Based on our experience, inclusion of 20 placebo- and 20 Semaglutide-treated subjects is suitable to perform the pilot study. We hypothesize a ≥10% decrease in global disease score as measured by NaF uptake in the heart and/or thoracic aorta, will be present after 30 weeks treatment. Will not be covered in primary publication. The results will be presented in a separate puplication.
Positive and Negative Symptom Scale 6 | 30 Weeks
  Positive and Negative Symptom Scale 6 (PANSS-6): PANSS-6 is an operationalized rating of positive and negative symptoms, in people with schizophrenia, which is sensitive to change. PANSS-6 is a shorter version of the original 30-item version. It is validated and translated into Danish and has proven a good level of inter-rater reliability when rated based on the Simplified Negative and Positive Symptoms Interview (SNAPSI). PANSS-6 interview will be performed at baseline, and after 15 and 30 weeks. Minimum score: 6. Maximum score 42. Higher scores indicate more severe symptoms. These results will be presented in the primary publication.
Impact of Weight on Quality of Life-Lite | 30 Weeks
  Impact of Weight on Quality of Life-Lite (IWQOL-Lite): IWQOL-Lite is a reliable and valid self-report measure for assessing weight-related QoL in people with schizophrenia. It provides a total score plus scores on five domains (physical function, self-esteem, sexual life, public distress, and work). IWQOL-Lite will be measured at baseline, and after 15 and 30 weeks. It consist of 31 items with scores in multiple domains. The score is transformed into 0-100 scale (100 being best quality of life). Will not be covered in primary publication.
Short Form Survey version 2 (SF-36v2) | 30 Weeks
  SF-36v2 is a well-researched, self-reported measure of health. It comprises 36 questions in 8 different domains. The survey will be applied in Danish, using the latest updated version 2 (SF-36v2). It will be measured at baseline, week 15 and week 30. Scoring of the health domain scales involves: (a) recoding item response values, (b) summing recoded response values for all items in a given scale to obtain the scale raw score, (c) transforming the scale raw score to a 0-100 score, (d) transforming the 0-100 score to a z score, and (e) transforming the scale z score to a T score (mean = 50, standard deviation = 10). In general, for individual respondents, T scores of 45 or greater indicate at least average overall functioning or well-being in the health domain or overall health dimension-physical or mental-being assessed, as compared to the U.S. general population. These results will be presented in the primary publication.
Medication Adherence Rating Scale | 30 Weeks
  Medication Adherence Rating Scale (MARS): MARS is a validated and reliable measure of adherence for psychoactive medication. MARS constitutes 10 items rating the medical adherence. MARS will be measured at baseline, and at weeks 5, 9, 15, 19, 23, 28 and 30. Total scores range from 0 (low likelihood of medication adherence) to 10 (high likelihood). These data will not be presented in the primary publication.
The Simple Physical Activity Questionnaire | 30 Weeks
  The Simple Physical Activity Questionnaire (SIMPAQ): SIMPAQ has shown good test-retest reliability and has been validated against measures from Actigraph accelerometers. SIMPAQ will be measured at baseline, and at weeks 5, 9, 15, 19, 23, 28 and 30. The 5-item SIMPAQ required people being interviewed to account for time spent in bed overnight, time sedentary, including napping, time spent walking, time spent exercising and time engaged in incidental activity, averaged over the past seven-day period. The sum of the hours recorded in the five SIMPAQ boxes should add to approximately 24-h. Will not be covered in primary publication.
EQ-5D-3L | 30 Weeks
  EQ-5D-3L is a widely applied instrument for the measurement and cost-benefit evaluation of health interventions. EQ-5D-3L will be measured at baseline, and at weeks 5, 9, 15, 19, 23, 28 and 30. EQ-5D-3L consists of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Within each dimension, there are three levels: no problems, some problems, and extreme problems. Patients are required to designate their health state by marking the box corresponding to the most relevant statement for each dimension. This choice yields a single-digit number representing the selected level for that dimension. These digits across the five dimensions can be assembled into a 5-digit number that characterizes the patient's overall health state. A total of 243 possible health states is defined in this way. A score of 11111 indicates the best health, while a score of 33333 reflects the poorest health. Will not be covered in primary publication.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Frystyk, Professor, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Biological material / biobank:
  Biological material will be stored in a research biobank to be analysed in the end of trial, hereby we can analyse all non-safety variables at the same lab with the same assays to minimize differences in lab technique and differences in assays.
  In addition biological material will also be collected and stored in a biobank for future unspecific research projects. Biological material will be stored in pseudo-anonymised form by ID-number in a biobank for 15 years, after which it will be destroyed. In case there is a need for further studies of biomaterial, application will again be made to the Science Ethics Committee.
Supporting Information: Study Protocol
Time Frame: 15 years
Access Criteria: In case there is a need for further studies of biomaterial, application will again be made to the Science Ethics Committee.

REFERENCES:
- [Derived] Ganeshalingam AA, Uhrenholt N, Arnfred S, Gaede P, During S, Stenager EN, Bunger N, Pedersen AK, Bilenberg N, Frystyk J. Semaglutide Treatment of Antipsychotic-Treated Patients With Schizophrenia, Prediabetes, and Obesity: The HISTORI Randomized Clinical Trial. JAMA Psychiatry. 2025 Nov 1;82(11):1065-1074. doi: 10.1001/jamapsychiatry.2025.2332. PMID 40900607
- [Derived] Ganeshalingam AA, Uhrenholt NG, Arnfred S, Gaede PH, Bilenberg N, Frystyk J. Home-based Intervention with Semaglutide Treatment of Neuroleptic-Related Prediabetes (HISTORI): protocol describing a prospective, randomised, placebo controlled and double-blinded multicentre trial. BMJ Open. 2024 Mar 18;14(3):e077173. doi: 10.1136/bmjopen-2023-077173. PMID 38503415

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-07-05): https://cdn.clinicaltrials.gov/large-docs/78/NCT05193578/SAP_003.pdf